CLINICAL TRIAL: NCT03080870
Title: JOY of ART - an Intervention Study for Older Adults and Their Family Caregivers
Brief Title: JOYof ART - an Intervention Study
Acronym: JOYofART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Eastern Finland (Other)
Collaborators: Kuopio Conservatory (Unknown); Kuopio University Hospital (Other); Savonia University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Tarja Välimäki, Principal Investigator, University of Eastern Finland
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: JOYof ART
Record Dates: First submitted 2017-02-21; First posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Quality of Life; Family Caregivers
Keywords: Art intervention; Quality of Life; Well-being; Physical performance; Family caregivers; Older adults
MeSH Terms: interventions — Reproductive Techniques, Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Art groups are held once a week, each with the duration of 60 minutes. They begin with a 45 minute art intervention and conclude with a 15 minute discussion. The art groups include music, dance and visual arts, which is psychologically, socially, and physically activating. Music has the main emphasis in art intervention. The preferences of the subjects are taken into consideration in art intervention. Art intervention is conducted by trained and experienced art pedagogues.
  Art intervention aims to revive previously learned art-related skills, to learn and enhance new skills, and to improve and intensify physiological, emotional, social, motoric, and cognitive abilities.
  Interventions: Other: Art
- Control (No Intervention): Baseline and follow-up measurements.

INTERVENTIONS:
Other: Art — Multicomponent art intervention
  Arms: Intervention

SUMMARY:
Music, dance and visual arts are suggested to support health and well-being of older people. Intervention studies, however, are scarce. JOY of ART study investigates the effects of multicomponent art intervention among older people and ther family caregivers.

DETAILED DESCRIPTION:
JOY of ART study investigates the effects of group based intervention including music, dance and visual arts. Art sessions are provided once a week in three months period each session takes 60 minutes. Eligible participants are recruited from the City of Kuopio, Finland, total 60 dyads, 30 to intervention group and 30 to control group. Health, physical performance and quality of life assessments are conducted at the baseline and in the end of the intervention. In addition, participants are contacted by phone and interviewed six months after the intervention has completed. For family caregivers qualitative interviews are conducted at the baseline and in the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* 65+ age, family caregiving dyad, ability to walk independently or assisted, home dwelling

Exclusion Criteria:

* severe dementia, severe aphasia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Mental Well-being assessed using the Warwick-Edinburgh Mental Well-being scale (WEMWBS) | Change in Mental Well-being from baseline until three month follow-up
  The Warwick-Edinburgh Mental Well-being scale (WEMWBS)

SECONDARY OUTCOMES:
Mobility and Balance assessed using Timed up & Go (TUG) | Change in Mobility and Balance from baseline until three month follow-up
  Timed up & Go (TUG)
Physical Performance assessed using Short Physical Performance Battery (SPPB) | Change in Physical Performance from baseline until three month follow-up
  Short Physical Performance Battery (SPPB)
Quality of Life assessed using EQ- 5D-5L | Change in Quality of Life from baseline until three month follow-up
  EQ- 5D-5L
Psychological Distress assessed using General Health Questionnaire (GHQ 12) | Change in Psychological Distress from baseline until three month follow-up
  General Health Questionnaire (GHQ 12)
Use of Social and Health Care Services assessed using Questionnaire | Change in use of Social and Health Care Service use from baseline until three month follow-up
  Questionnaire on Social and Health Care service use

CONTACTS AND LOCATIONS:
Locations (1):
- University of Eastern Finland, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pohjola H, Vaajoki A, Valimaki T. Art intervention among Finnish older people and their caregivers: Experiences of art pedagogies. Health Soc Care Community. 2020 Sep;28(5):1780-1786. doi: 10.1111/hsc.13003. Epub 2020 Apr 26. PMID 32337789